CLINICAL TRIAL: NCT05670236
Title: Effect of Knee Pain on Walking Biomechanics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Daniel Corrigan, Assistant Professor, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 32283
Record Dates: First submitted 2022-11-29; First posted 2023-01-04 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Gait; Pain; Osteoarthritis; Biomechanics
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Arm 1: Clinically defined unilateral symptomatic knee osteoarthritis;
  Arm 2: Healthy Controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Knee Osteoarthritis (Experimental): Individuals with clinically defined unilateral symptomatic knee osteoarthritis.
  Interventions: Drug: Lidocaine Hydrochloride
- Healthy (No Intervention): Individuals who serve as healthy controls.

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — 10 mL of 1% lidocaine hydrochloride for each intraarticular knee injection
  Arms: Knee Osteoarthritis

SUMMARY:
The goal of this study is to determine if pain in one knee influences loading of the other knee during different types of walking. The main questions it aims to answer are:

* How does unilateral knee pain affect contralateral knee joint loading during different types of walking?
* Does movement and loading change at the hips, knees, and ankles during prolonged walking in persons with painful knee osteoarthritis?

Participants will:

* Fill out questionnaires/surveys
* Complete clinical examinations
* Walking on a treadmill under different types of walking conditions
* Receive two knee injections For comparison purposes, researchers will also enroll healthy participants.

DETAILED DESCRIPTION:
This study will evaluate the effects of unilateral knee pain on contralateral knee joint loading during different types of walking. Thirty adults with unilateral symptomatic knee osteoarthritis will complete four, 1.5-hour study visits. The first and third visits will include level, inclined, and declined walking at comfortable, fast, and slow speeds. The second and fourth visits will include a 30-minute walk. There will be at least two days between visits. The only difference between each pair of visits is that one visit will involve walking with unilateral knee pain (painful walking) and the other visit will involve walking without unilateral knee pain (nonpainful walking). Individuals will be recruited based on the presence of unilateral knee pain so the painful walking will be representative of their typical walking. For the visits with nonpainful walking, the third and fourth visits, pain will be alleviated by performing an intraarticular injection with a local anesthetic (lidocaine hydrochloride). All walking will be performed in a three-dimensional motion capture environment on a split-belt treadmill that is instrumented with force plates.

A cohort of 30 healthy individuals will complete the same walking conditions at two, 1.5-hour study visits. The healthy control group will not receive intraarticular knee injections. The purpose of this cohort is to better understand how walking mechanics in individuals with unilateral knee osteoarthritis compare to similar individuals without knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria for Knee Osteoarthritis Arm:

* At least 45 years old
* Unilateral knee pain with walking that averages at least 3 out of 10 on a numeric pain rating scale
* Unilateral knee stiffness that lasts less than 30 minutes after periods of inactivity
* Unilateral symptoms on most days for at least the past 3 months

Exclusion Criteria for Knee Osteoarthritis Arm:

* History of knee replacement surgery
* Opiate use within the past 3 months
* Narcotic use within the past 3 months
* Known medical condition that affects walking mechanics, besides knee osteoarthritis
* Known medical condition that affects pain perception
* Inability to walk for 30 minutes without using an assistive device
* Body weight greater than 300 pounds
* Known allergy to adhesives
* High risk for a cardiovascular event
* Currently pregnant
* Anticoagulant use within the past 3 months
* Intraarticular knee injection within the past 3 months
* Known history of hypersensitivity to local anesthetics of the amide type
* History of lower body pain or injury, besides knee osteoarthritis, within the past 6 months

Inclusion Criteria for Healthy Arm:

* At least 45 years old
* No lower body pain or injury within the past 6 months

Exclusion Criteria for Healthy Arm:

* History of knee replacement surgery
* Opiate use within the past 3 months
* Narcotic use within the past 3 months
* Known medical condition that affects walking mechanics
* Known medical condition that affects pain perception
* Inability to walk for 30 minutes without using an assistive device
* Body weight greater than 300 pounds
* Known allergy to adhesives
* High risk for a cardiovascular event
* Currently pregnant

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Corrigan, DPT, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Knee Osteoarthritis | Healthy
Started (Baseline Testing) | 30 | 25
Completed (Entire Protocol) | 23 | 24
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Knee Osteoarthritis | Healthy | Total
Number analyzed (Participants) | 30 | 25 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.5) | 57.9 (7.8) | 60.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 24 | 20 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 25 | 55
Height [Mean (Standard Deviation); unit: cm] | 169.2 (10.0) | 171.1 (8.0) | 170.1 (9.1)
Weight [Mean (Standard Deviation); unit: kg] | 81.7 (20.7) | 77.5 (17.7) | 79.8 (19.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Medial Knee Contact Forces During Walking
Description: Contact forces estimated with musculoskeletal modeling
Time Frame: Change from before treatment (approximately 1 week prior to the injection visit) to 30 minutes after treatment (the injection).
Population: The healthy control group did not receive a treatment. Therefore, no change was expected or measured.
Measure: Mean (Standard Deviation); unit: bodyweights
Arm/Group | Knee Osteoarthritis | Healthy
Number analyzed (Participants) | 24 | 0
bodyweights | -0.04 (0.02) |

2. Primary Outcome: Change in Lateral Knee Contact Forces During Walking
Description: Contact forces estimated with musculoskeletal modeling
Time Frame: as for outcome 1
Population: The healthy control group did not receive a treatment. Therefore, no change was expected or measured.
Measure: Mean (Standard Deviation); unit: bodyweights
Arm/Group | Knee Osteoarthritis | Healthy
Number analyzed (Participants) | 24 | 0
bodyweights | 0.02 (0.03) |

3. Primary Outcome: Change in Patellofemoral Knee Contact Forces During Walking
Description: Contact forces estimated with musculoskeletal modeling
Time Frame: as for outcome 1
Population: The healthy control group did not receive a treatment. Therefore, no change was expected or measured.
Measure: Mean (Standard Deviation); unit: bodyweights
Arm/Group | Knee Osteoarthritis | Healthy
Number analyzed (Participants) | 24 | 0
bodyweights | -0.01 (0.01) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each study visit. All study visits occurred within a one-month period.
Arm/Group | Knee Osteoarthritis | Healthy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT05670236/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT05670236/ICF_001.pdf